CLINICAL TRIAL: NCT04397679
Title: Treatment of Adults with Newly Diagnosed Glioblastoma with Partial Brain Radiation Therapy Plus Temozolomide and Chloroquine Followed by Tumor Treating Fields Plus Temozolomide and Chloroquine -- a Pilot Study
Brief Title: Partial Brain RT, Temozolomide, Chloroquine, and TTF Therapy for the Treatment of Newly Diagnosed Glioblastoma
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: slow accrual
Sponsor: Barbara Ann Karmanos Cancer Institute (Other)
Responsible Party: Principal Investigator, Michael Dominello, Principal Investigator, Barbara Ann Karmanos Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2018-148
Record Dates: First submitted 2020-05-18; First posted 2020-05-21 (Actual); Last update posted 2025-01-15 (Actual); Status verified 2025-01

CONDITIONS: Glioblastoma; Gliosarcoma
MeSH Terms: conditions — Glioblastoma; Gliosarcoma | interventions — Radiotherapy, Conformal; Radiation; Radiotherapy, Intensity-Modulated; Temozolomide; Chloroquine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Treatment (radiation therapy, temozolomide, chloroquine, TTF) (Experimental): Patients undergo 30 fractions of 3D CRT or Intensity-modulated radiation therapy (IMRT) and receive temozolomide by mouth (PO) and chloroquine PO daily from day 1 for the duration of radiation therapy up to day 49. Treatment continues in the absence of disease progression or unacceptable toxicity.
  ADJUVANT TREATMENT: Beginning 4 weeks after the last day of radiation therapy, patients receive temozolomide PO QD on days 1-5 and chloroquine PO daily on days 1-28. Treatment repeats every 28 days for up to 6 cycles in the absence of disease progression or unacceptable toxicity. Patients demonstrating continued benefit may continue to receive temozolomide and chloroquine for up to 12 cycles. Patients also undergo TTF therapy over 18 hours or longer per day.
  Interventions: Radiation: 3-Dimensional Conformal Radiation Therapy; Radiation: Intensity-Modulated Radiation Therapy (IMRT); Drug: Temozolomide; Drug: Chloroquine; Procedure: Tumor Treating Fields Therapy (TTF)

INTERVENTIONS:
Radiation: 3-Dimensional Conformal Radiation Therapy — Undergo 3D CRT
  Other Names: 3-dimensional radiation therapy; 3D CONFORMAL RADIATION THERAPY; 3D CRT; 3D-CRT; Conformal Therapy; Radiation Conformal Therapy; Radiation; 3D Conformal
Radiation: Intensity-Modulated Radiation Therapy (IMRT) — Undergo IMRT
  Other Names: IMRT; Intensity Modulated RT; INTENSITY-MODULATED RADIATION THERAPY; Intensity-Modulated Radiotherapy; Radiation
Drug: Temozolomide — Given PO
  Other Names: 3,4-dihydro-3-methyl-4-oxoimidazo[5,1-d]-1,2,3,5-tetrazine-8-carboxamide, 362856; 8-carbamoyl-3-methylimidazo[5,1-d]-1,2,3,5-tetrazin-4(3H)-one, 85622-93-1, CCRG-81045; imidazo[5,1-d]-1,2,3,5-tetrazine-8-carboxamide, 3; 4-dihydro-3-methyl-4-oxo-, Imidazo[5,1-d]; 1,2,3,5-tetrazine-8-carboxamide; 3, 4-dihydro-3-methyl-4-oxo-, M & B 39831, M and B 39831; Methazolastone; RP-46161; SCH 52365; Temcad; Temodal; Temomedac; TMZ
Drug: Chloroquine — Given PO
  Other Names: 54-05-7
Procedure: Tumor Treating Fields Therapy (TTF) — Undergo TTF
  Other Names: Alternating Electric Field Therapy; TTF; TTFields

SUMMARY:
This trial studies the side effects of partial brain radiation therapy, temozolomide, chloroquine, and tumor treating fields therapy for the treatment of newly diagnosed glioblastoma. Radiation therapy uses high energy x-rays to kill tumor cells and shrink tumors. Chemotherapy drugs, such as temozolomide, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Chloroquine is normally used to treat strains of malaria and prior preclinical and clinical data suggests that it may increase the efficacy of both radiation and tumor treating fields therapy. Tumor treating fields therapy uses electric fields tuned to specific frequencies to disrupt cell division, inhibiting tumor growth and potentially causing cancer cells to die. The purpose of this study is to determine the safety of partial brain radiation therapy, temozolomide, chloroquine, and tumor treating fields therapy in patients with gliobastoma

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine the safety of partial brain radiation therapy plus temozolomide and chloroquine followed by tumor treating fields (TTFs) plus temozolomide and chloroquine, specifically grade 3 or higher dermatitis within the first 3 months of the adjuvant therapy phase.

SECONDARY OBJECTIVE:

I. To measure treatment effect via advanced magnetic resonance imaging (MRI) and alpha-[11C]methyl-L-tryptophan (AMT)-positron emission tomography (PET).

OUTLINE:

Patients undergo 30 fractions of 3-dimensional conformal radiation therapy (3D CRT) or intensity-modulated radiation therapy (IMRT) and receive temozolomide orally (PO) and chloroquine PO daily from day 1 for the duration of radiation therapy up to day 49. Treatment continues in the absence of disease progression or unacceptable toxicity.

ADJUVANT TREATMENT: Beginning 4 weeks after the last day of radiation therapy, patients receive temozolomide PO once daily (QD) on days 1-5 and chloroquine PO daily on days 1-28. Treatment repeats every 28 days for up to 6 cycles in the absence of disease progression or unacceptable toxicity. Patients demonstrating continued benefit may continue to receive temozolomide and chloroquine for up to 12 cycles. Patients also undergo TTF therapy over 18 hours or longer per day.

After completion of study treatment, patients are followed up monthly for 3 months.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed newly diagnosed grade IV glioma (gliosarcoma allowed)
* The subject must have recovered from the effects of surgery, postoperative infection, and other complications before enrollment. Post-operative unenhanced and contrast-enhanced MRI scan should be done within 72 hours after surgery. If it is not obtained within 72 hours post-resection, then an MRI obtained at least 2 weeks (or longer) after surgery is required
* Karnofsky performance status >= 70%
* Absolute neutrophil count >= 1,500/mm^3 (=< 21 days prior to registration)
* Platelets >= 100,000/mm^3 (=< 21 days prior to registration)
* Hemoglobin (Hgb) >= 9.0 g/dL (Note: The use of transfusion or other intervention to achieve Hgb >= 9.0 g/dL is acceptable.) (=< 21 days prior to registration)
* Calculated creatinine clearance >= 30 mL/min by Cockcroft-Gault formula (=< 21 days prior to registration)
* Total bilirubin =< 1.5 times upper limit of normal (ULN) (=< 21 days prior to registration)
* Aspartate aminotransferase (AST)(serum glutamic-oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT)(serum glutamate pyruvate transaminase [SGPT]) =< 1.5 times upper limit of normal (ULN) (=< 21 days prior to registration)
* Female subjects of childbearing potential (i.e., those who are not postmenopausal for at least 1 year or surgically sterile by bilateral tubal ligation, bilateral oophorectomy or hysterectomy) and their male partners should practice at least one of the methods of birth control listed below during study entry, for the entire duration of the study and for at least 6 months after treatment with temozolomide and chloroquine:

  * A vasectomized male subject or a vasectomized partner of a female subject; hormonal contraceptives (oral, parenteral, or transdermal) for at least 3 months prior to study drug administration; intrauterine device (females); double-barrier method (condoms, contraceptive sponge, diaphragm or vaginal ring with spermicidal jellies or cream)
* Female subjects of child-bearing potential must have a negative pregnancy test (urine or serum) within 3 days of registration
* Must voluntarily sign and date informed consent form for study participation, approved by an Independent Ethics Committee (IEC)/Institutional Review Board (IRB), prior to the initiation of any screening or study-specific procedures

Exclusion Criteria:

* Gliomatosis cerebri (a diffuse glioma [usually astrocytic] growth pattern consisting of exceptionally extensive infiltration of a large region of the central nervous system, with involvement of at least 3 cerebral lobes, usually with bilateral involvement of the cerebral hemispheres and/or deep grey matter, and frequent extension to the brain stem, cerebellum, and even the spinal cord.)
* Recurrent glioblastoma (GBM)
* Metastatic GBM
* Infratentorial tumor
* Prior chemotherapy or radiosensitizers for cancers of the head and neck region; note that prior chemotherapy for a different cancer is allowable, except prior temozolomide. Implanted carmustine (BCNU) wafer is allowed
* Prior radiotherapy to the head or neck (except for T1 glottic cancer or nonmelanomatous skin cancer), resulting in overlap of radiation fields
* Any prior therapy for glioblastoma besides surgery (intra-operative techniques to guide resection and experimental imaging techniques are allowed). BCNU wafer is allowed
* Prior invasive malignancy (except for non-melanomatous skin cancer; carcinoma in situ (CIS) of the breast, CIS oral cavity, or CIS cervix, T1 glottic cancer) unless disease free for >= 5 years
* Prior, concomitant, or planned concomitant treatment with bevacizumab, carmustine implant (Gliadel) wafers or other intratumoral or intracavitary anti-neoplastic therapy, or other experimental therapeutics intended to treat the tumor; the exceptions are diagnostic and operative guides to improve extent of resection or imaging studies, quality of life, biomarker, or epidemiological studies
* History of hypersensitivity to temozolomide or excipients
* Known glucose-6-phosphate dehydrogenase (G6PD) deficiency
* Lactating or pregnant female
* Severe, active, co-morbidity defined as follows:

  * Moderate or severe hepatic impairment (Child-Pugh category B or higher [score of 7 or higher ]); unstable angina and/or congestive heart failure within the last 6 months; transmural myocardial infarction within the last 6 months; evidence of recent myocardial infarction or ischemia by the findings of S-T elevations of >= 2 mm using the analysis of an electrocardiogram (EKG) performed within 14 days prior to enrollment; New York Heart Association grade II or greater congestive heart failure requiring hospitalization within 12 months prior to enrollment
* History of stroke, cerebral vascular accident (CVA), or transient ischemic attack within 6 months (except if intra- or post-operative); serious and inadequately controlled cardiac arrhythmia; acute bacterial or fungal infection requiring intravenous antibiotics at the time of enrollment; chronic obstructive pulmonary disease exacerbation or other respiratory illness requiring hospitalization or precluding study therapy at the time of enrollment; uncontrolled human immunodeficiency virus (HIV) with CD4 count < 200; note, however, that HIV testing is not required for entry into this protocol
* Any other major medical illnesses or psychiatric impairments that in the investigator's opinion will prevent administration or completion of protocol therapy
* Subjects treated on any other therapeutic clinical protocols within 30 days prior to study entry or during participation in the study, except intra-operative therapy to guide resection or experimental imaging without therapeutic intent
* Inability to undergo contrast-enhanced MRI scans
* Presence of implanted pacemaker, programmable shunts, defibrillator, deep brain stimulator, or other implanted electronic devices in the brain
* Documented clinically significant arrhythmia or severe ischemic heart disease
* Patients with underlying ocular disorders, including but not limited to: maculopathy, macular degeneration, and retinopathy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2021-08-12 (Actual); Primary Completion 2024-05-14 (Actual); Study Completion 2024-05-14 (Actual)

PRIMARY OUTCOMES:
Proportion of patients who develop a specific acute toxicity (dermatitis) | First 3 months of adjuvant therapy phase
  Will summarize dermatitis status

SECONDARY OUTCOMES:
Incidence of adverse events | First 3 months of adjuvant therapy phase
  Will detail the safety profile and measure (via magnetic resonance imaging and positron emission tomography scans) the uptake and retention of alpha-[11C]methyl-L-tryptophan.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Dominello, M.D., Principal Investigator — Barbara Ann Karmanos Institute
Locations (1):
- Barbara Ann Karmanos Cancer Institute, Detroit, Michigan, United States